CLINICAL TRIAL: NCT00958958
Title: Brazilian Intervention to Increase Evidence Usage in Practice - Acute Coronary Syndromes
Acronym: BRIDGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IEP012009
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; randomized cluster trial; quality improvement
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quality improvement program (Other): There are multifaceted Interventions for the clinic hospital team Including
  1. Distribution of educational materials
  2. Case manager
  3. Reminders
  4. Practical training
  Interventions: Other: multifaceted strategy
- Hospital standard treatment (No Intervention): Hospital standard treatment

INTERVENTIONS:
Other: multifaceted strategy — There are multifaceted Interventions Including
  1. Distribution of educational materials: distribution of published or printed recommendations for clinical care.
  2. Case manager: Use of a trained person who works in the hospital and will be responsible to assure that all interventions were used
  3. Reminders
  4. Practical training
  Arms: Quality improvement program

SUMMARY:
Phase 1: An observational study (registry) will be conducted which will objectively document the ACS clinical practice in Brazilian public hospitals, and identify the important barriers for the evidence usage incorporation in the clinical practice.

Phase 2: A Cluster randomized clinical trial in which public hospital will be randomized to receive or not a multifaceted strategy in order to increase evidence based therapy in clinical practice.

DETAILED DESCRIPTION:
STUDY POPULATION:

Patients with thoracic pain who the emergency department physician suspects of ACS and plans start a treatment for this issue; It will be excluded patients transferred of others institutions with 12 hours of symptoms.

PROGRAM:

There are multifaceted Interventions Including

1. Distribution of educational materials
2. Case manager: Use of a trained person who works in the hospital and will be responsible to assure that all interventions were used
3. Reminders: specific information that is designed or intended to prompt a health professional to recall information (patient bracelets, labels, posters, pocket cards, checklists).
4. Practical training

ENDPOINTS:

Phase 1 Primary outcome; patient who've received interventions based on evidence proportion informed by the indicators; Phase 2

Primary outcome:

Increase of prescription of evidence based treatment in clinical practice Secondary outcome Total mortality and major cardiovascular events

ELIGIBILITY:
Patient Eligibility criteria

Inclusion Criteria:

* Patients with thoracic pain who the emergency department physician suspects of ACS and plans start a treatment for this issue

Exclusion Criteria:

* Patients transferred from others institutions within 12 hours of the symptoms

Cluster Eligibility Criteria

* National Public Hospitals with emergency department. A cluster can be one hospital with emergency department, or 2 or more hospitals (for example: 1 emergency hospital and 1 general hospital which receive the patients to perform PCI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2010-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Phase 1: patient who've received interventions based on evidence proportion informed by the indicators | 9 months
Phase 2: increase of prescription of evidence based treatment in clinical practice | 6 months

SECONDARY OUTCOMES:
Total mortality and major cardiovascular events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Otávio Berwanger, PhD, Principal Investigator — Hospital do Coracao
Locations (1):
- Hospital do Coração, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Berwanger O, Guimaraes HP, Laranjeira LN, Cavalcanti AB, Kodama AA, Zazula AD, Santucci EV, Victor E, Tenuta M, Carvalho V, Mira VL, Pieper KS, Weber B, Mota LH, Peterson ED, Lopes RD; Bridge-Acs Investigators. Effect of a multifaceted intervention on use of evidence-based therapies in patients with acute coronary syndromes in Brazil: the BRIDGE-ACS randomized trial. JAMA. 2012 May 16;307(19):2041-9. doi: 10.1001/jama.2012.413. PMID 22665103
- [Derived] Berwanger O, Guimaraes HP, Laranjeira LN, Cavalcanti AB, Kodama A, Zazula AD, Santucci E, Victor E, Flato UA, Tenuta M, Carvalho V, Mira VL, Pieper KS, Mota LH, Peterson ED, Lopes RD; BRIDGE-ACS. A multifaceted intervention to narrow the evidence-based gap in the treatment of acute coronary syndromes: rationale and design of the Brazilian Intervention to Increase Evidence Usage in Acute Coronary Syndromes (BRIDGE-ACS) cluster-randomized trial. Am Heart J. 2012 Mar;163(3):323-29, 329.e1. doi: 10.1016/j.ahj.2012.02.004. PMID 22424001